CLINICAL TRIAL: NCT03022695
Title: Treatment of Breast Fibroadenoma With High Intensity Focused Ultrasound (HIFU)
Acronym: HIFU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Theraclion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIFU 1.0
Record Dates: First submitted 2015-07-01; First posted 2017-01-16 (Estimated); Last update posted 2024-07-22 (Actual); Status verified 2015-06

CONDITIONS: Breast Fibroadenoma
MeSH Terms: conditions — Fibroadenoma

ARMS (1):
- Treatment with high-intensity focused ultrasound (Experimental)
  Interventions: Device: High Intensity Focused Ultrasound

INTERVENTIONS:
Device: High Intensity Focused Ultrasound

SUMMARY:
This is a monocenter, open-label, uncontrolled study in accordance with §23b MPG to evaluate the efficacy of the HIFU-treatment of fibroadenoma using the TH-One device.

ELIGIBILITY:
Inclusion Criteria:

* Female patients 18 years or older with at least one diagnosed breast fibroadenoma. Diagnosis of fibroadenoma must be based on:
* clinical examination,
* women ≤ 40 years of age: ultrasound image alone; women > 40 years of age: ultrasound image and mammogram,
* histological confirmation of fibroadenoma of the breast. Patient's fibroadenoma size as determined by ultrasound imaging: the longest diameter is limited to 25 mm. Women of childbearing potential must have a negative urine pregnancy test within 72 hours prior to HIFU treatment. Patient must be able to understand the nature and the extent of the study and the procedures required and be willing and able to complete the screening and study procedures. Patient must give written informed consent (personally signed and dated) before completing any study-related procedure.

Exclusion Criteria:

* Patient who is pregnant or breast-feeding.
* Patient with history of ipsilateral breast cancer within 5 years prior to study inclusion or radio therapy to the target breast within 5 years prior to study inclusion.
* Patient with implant on the treated breast.
* Patient with target fibroadenoma pre-treated by cryoablation or interstitial laser therapy within 12 month before recruiting for HIFU.
* Patient's fibroadenoma not clearly visible on the ultrasound images (in B mode) at the inclusion visit. Patient participating in other studies using drugs or medical devices within 3 months prior to study inclusion or during study participation including the follow-up period.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2013-10; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
The efficacy is assessed by a reduction in volume of the fibroadenoma at baseline, 6 months and at 12 months after the HIFU on the ultrasonography. | Baseline, 6 months, 12 months
  A reduction in volume of > 65% compared to baseline, or a total regression of the fibroadenoma will be taken as effective treatment. The results will be analyzed descriptively

SECONDARY OUTCOMES:
Energy setting to obtain reduction in volume or total regression of the fibroadenoma at 12 months follow-up | 1 year
Lack of palpable lesion | 2 years
Pain free if pain at baseline (pain related to the fibroadenoma) | 1 year
Gland vascularisation (compared to baseline) power Doppler at day 7, month 6 and 12 after the HIFU session | Day 7, month 6, month 12
Pain during the HIFU session using a Visual Analog Pain Scale | 0 month
Histological outcome through core needle biopsy after 12 month | 1 year
Quality and ease of use of breast immobilization | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Department for Women's Health, Tübingen, Germany